CLINICAL TRIAL: NCT00653757
Title: Phase I/II Study of Radioimmunoguided Intensity Modulated Radiotherapy (IMRT) for Prostate Cancer
Brief Title: Intensity-Modulated Radiation Therapy in Treating Patients With Stage I, Stage II, Stage III, or Stage IV Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven E Schild, M.D., Mayo Clinic Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000588847; P30CA015083 (NIH); 390-02 (Other: Mayo Clinic Cancer Center); 390-02 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-04-04; First posted 2008-04-07 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; Leuprolide; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: goserelin acetate
Drug: leuprolide acetate
Radiation: image-guided radiation therapy
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Using scintigraphy to plan specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I/II trial is studying the side effects and best way to give intensity-modulated radiation therapy and to see how well it works in treating patients with stage I, stage II, stage III, or stage IV prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the feasibility of radioimmunoguided intensity-modulated radiotherapy (IMRT) for stage I-IV prostate cancer.
* To determine the toxicity and tolerance of this regimen in these patients.
* To determine the tumor response based on physical examination and serial measurements of the serum prostate-specific antigen (PSA) levels in these patients.
* To determine the outcome of patients treated on this study with radioimmunoguided IMRT compared to 2 control groups of patients treated at Mayo Scottsdale Clinic (MSC).

OUTLINE: Patients undergo radioimmunoguided intensity-modulated radiotherapy once daily, 5 days a week for 8½ weeks. Beginning the last week of radiotherapy, some patients receive leuprolide acetate intramuscularly every 3-4 months or goserelin subcutaneously every 3 months for 6 months, 12 months, or until disease progression.

After completion of study treatment, patients are followed every 3-4 months for 1 year, every 6 months for 4 years and annually thereafter

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed prostate cancer

  * Stage I-IV disease (T1-4, N0-1, M0)
* No evidence of distant metastases (M0) on physical examination or bone scan

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Hemoglobin ≥ 10.0 g/dL
* WBC ≥ 3,000/mcL
* Platelet count ≥ 90,000/mm
* AST < 2 times the upper limit of normal
* No allergy to leuprolide acetate or goserelin

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-03; Primary Completion 2006-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Toxicity
Survival rates
Freedom from biochemical relapse rates
Local control rates
Distant failure rates
Biochemical freedom from failure rates
Comparison of outcomes to patients treated with conventional radiotherapy and intensity-modulated radiotherapy without radioimmunoguidance

SECONDARY OUTCOMES:
Obstructive urinary symptoms
Sexual health as assessed by inventory questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Schild, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States